CLINICAL TRIAL: NCT02983773
Title: Marijuana's Impact on Alcohol Motivation and Consumption
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jane Metrik, Associate Professor (research), Brown University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1511001372; R01AA024091 (NIH)
Record Dates: First submitted 2016-11-15; First posted 2016-12-06 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Alcohol Drinking; Marijuana
MeSH Terms: conditions — Alcohol Drinking; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High THC dose (Experimental): 1 marijuana cigarette (7.2% THC)
  Interventions: Drug: THC 7.2%
- Low THC dose (Experimental): 1 marijuana cigarette (3.0% THC)
  Interventions: Drug: THC 3.0%
- Placebo (Placebo Comparator): Placebo marijuana cigarette
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THC 7.2% — 1 smoked marijuana cigarette with 7.2% THC
  Arms: High THC dose
Drug: THC 3.0% — 1 smoked marijuana cigarette with 3.0% THC
  Arms: Low THC dose
Drug: Placebo — 1 smoked placebo marijuana cigarette
  Arms: Placebo

SUMMARY:
This laboratory study will employ a repeated measures experimental design to examine the effect of high (7.2% THC) and moderate (3% THC) dose of marijuana, relative to placebo, on alcohol craving and on behavioral economic measure of alcohol demand after exposure to alcohol cues, and on subsequent drinking in an alcohol choice task in which participants choose either to drink or receive monetary reinforcement for drinks not consume. The study will recruit 173 non-treatment seeking heavy episodic alcohol drinkers who smoke marijuana at least twice weekly.

DETAILED DESCRIPTION:
This laboratory study will employ a repeated measures experimental design to examine the effect of high (7.2% THC) and moderate (3.0% THC) dose of marijuana, relative to placebo, on alcohol craving and on behavioral economic measure of alcohol demand after exposure to alcohol cues, and on subsequent drinking in an alcohol choice task in which participants choose either to drink or receive monetary reinforcement for drinks not consumed. Moderators of the marijuana's effects on alcohol-related dependent variables will be tested: DSM5 alcohol use disorder severity, affective vulnerability, trait impulsivity, and working memory functioning. Several empirically-determined mechanisms that may explain why marijuana may increase risk of alcohol relapse and help maintain heavy drinking will be tested as mediators of marijuana's effects on alcohol. The study will recruit 173 non-treatment seeking heavy episodic alcohol drinkers who smoke marijuana at least twice weekly to obtain the final sample of 150 with complete data (15% of attrition). Participants will be tested at a baseline session and during three experimental sessions. Investigators will collect blood samples for analysis of cannabinoid plasma levels and to examine marijuana-induced changes in hormones and other biomarkers potentially related to appetite, inflammation and stress. Collection of these biomarkers would allow for a greater understanding about the mechanisms whereby marijuana may acutely increase alcohol motivation and use. The findings will inform researchers and clinicians about how marijuana acutely increases alcohol craving and consumption. The strategy of this proposal is to use the most comprehensive controlled test characterizing marijuana's putative effects on alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 44
* English-speaking
* marijuana smoking in past month
* report of current heavy episodic (binge) drinking
* in good physical health and weighing < 250 lbs
* zero breath alcohol at each visit

Exclusion Criteria:

* history of seizures
* smoking >20 tobacco cigarettes per day
* positive pregnancy test
* nursing
* positive urine toxicology screen for drugs other than cannabis
* interest to quit or receive treatment for marijuana or alcohol use
* meeting criteria for a current affective disorder (depression, or mania, panic disorder, and having psychotic symptoms as assessed by the SCID)

Ages: 21 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
change in alcohol craving | T1: pre-smoking (-45 minutes) and post smoking at 20 (T2), 55 (T3), and 70 (T4) minutes for a total of two hours during the experimental session
  Alcohol Craving Questionnaire-Short Form-Revised (ACQ-SF-R)

SECONDARY OUTCOMES:
change in alcohol demand measured with Alcohol Purchase Task-State Version (APT-SV) | T1: pre-smoking (-45 minutes) and post smoking at 55 (T2) and 70 (T3) minutes for a total of two hours during the experimental session
  Alcohol demand curve is generated by estimating alcohol consumption (number of drinks) over the course of escalating prices.
number of alcohol beverages consumed | post-smoking during two-hour alcohol choice task during the experimental session

CONTACTS AND LOCATIONS:
Overall Officials: Jane Metrik, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

DOCUMENTS (1):
  • Informed Consent Form (2020-06-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT02983773/ICF_000.pdf